CLINICAL TRIAL: NCT01281696
Title: A Phase II Study of Bevacizumab With Etoposide and Cisplatin in Breast Cancer Patients With Brain and/or Leptomeningeal Metastasis
Brief Title: Bevacizumab With Etoposide and Cisplatin in Breast Cancer Patients With Brain and/or Leptomeningeal Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Taichung Veterans General Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201010077M
Record Dates: First submitted 2010-12-24; First posted 2011-01-24 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Breast Neoplasms; Leptomeningeal Metastasis; Brain Metastases
Keywords: Breast cancer; CNS metastasis; Brain metastasis; Leptomeningeal metastasis; Bevacizumab; Etoposide; Cisplatin
MeSH Terms: conditions — Breast Neoplasms; Meningeal Carcinomatosis; Brain Neoplasms | interventions — Bevacizumab; Etoposide; Cisplatin; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab, etoposide, cisplatin (BEEP) (Experimental)
  Interventions: Drug: Bevacizumab, etoposide, cisplatin; Drug: Intrathecal methotrexate

INTERVENTIONS:
Drug: Bevacizumab, etoposide, cisplatin — Bevacizumab (15mg/kg) on D1, etoposide (70mg/m2) on D2-D4, cisplatin (70mg/m2) on D2; 21 days a cycle, for a maximum of 6 cycles
  Other Names: Bevacizumab (Avastin)
Drug: Intrathecal methotrexate — Additional intrathecal methotrexate only given in patients with leptomeningeal metastasis
  Other Names: Methotrexate

SUMMARY:
The main purpose of this study is to investigate the efficacy of bevacizumab, etoposide and cisplatin in treating breast cancer patients with central nervous system metastasis (including brain parenchymal and leptomeningeal metastasis).

DETAILED DESCRIPTION:
Brain metastases are increasingly important causes of morbidity and mortality in breast cancer patients. Whole brain radiotherapy (WBRT) and surgery remains the standard treatment for brain metastases. However, the median overall survival after brain and leptomeningeal metastasis were only 8.5 months and 16 weeks respectively There is lack of standard treatment for brain metastasis progression post WBRT. Chemotherapy was considered mostly poor for treatment response because of the blood brain barrier. However, this has been questioned because tumor can disrupt the normal function of blood brain barrier. For example, etoposide and cisplatin had been used for treatment for breast cancer patients with brain metastasis. The overall response rate of central nervous system (CNS) was 39 %, disease control rate was 60%, although the median overall survival was 31 weeks only. The role of targeted therapies is actively being assessed. Recently, a phase II study of lapatinib in patients with brain metastases from HER2-positive breast cancer showed that CNS objective response rates were 6% to lapatinib monotherapy and 20% to lapatinib plus capecitabine. Although the result is promising, the treatment population is limited in the HER2 overexpression breast cancer.

Bevacizumab, an anti-angiogenic agent, has been approved to combine with several chemotherapy agents in breast, lung and colon cancer. It was once considered contraindicated in patients with brain metastases due to the possibility of intracranial bleeding. However, two studies involving the use of bevacizumab for treating brain metastatic tumors of non-squamous or peripherally located squamous lung cancer showed no report of brain hemorrhage. In addition, bevacizumab has been approved to treat primary brain aggressive tumors recently.

In the institution, the investigators treated three breast cancer patients with multiple brain metastases using bevacizumab plus etoposide and cisplatin (B-EP). All of them have been treated for at least two lines of chemotherapy before brain metastases occurred. All of them received WBRT for brain metastases and one of them also received craniotomy with brain tumor resection plus local stereotactic radiosurgery. The follow up magnetic resonance imaging (MRI) had revealed recurrent metastatic brain tumors in one patients, and recurrence of leptomeningeal metastasis in another two patients. One patient who has multiple brain parenchyma metastases showed objective response on MRI after two cycle of B-EP treatment, and remained progression free for more than 5 months. The other two patients with leptomeningeal metastasis had intrathecal and intraventricular (via Ommaya reservoir) methotrexate treatment for more than eight doses. They were near stupor before B-EP treatment. Both had best clinical response of full recovery of consciousness and absence of cancer cells in cerebrospinal fluid. One survived eight months after the diagnosis leptomeningeal metastasis, and the other two were still alive six months after the diagnosis of leptomeningeal metastasis .

Dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) has been used in various studies for evaluation of anti-angiogenic condition. In breast cancer, DCE-MRI has been used as an early predictive marker for response. Glioblastoma patients have also been evaluated with DCE-MRI to determine reduction of vessel permeability after bevacizumab treatment.

Proton magnetic resonance spectroscopy (1H-MRS) has been used to different benign brain tumors from malignant ones. The utilization of 1H-MRS, especially in human brain tumors, coupled to both routine MRI and functional MRI techniques provides greater information concerning tumor grading and extension and characterization of the normal surrounding tissue than what is possible with any other imaging technique alone. To analyze proton spectroscopy before and after bevacizumab may give us further information about the mechanism of B-EP on CNS metastasis.

Therefore, the investigators propose to conduct a phase II clinical trial to test the efficacy of B-EP regimen in breast cancer patients with CNS metastasis along with brain DCE-MRI to demonstrate the antiangiogenesis efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. A histological confirmed invasive breast cancer
2. Patient with at least one measurable brain metastatic tumor (≧10mm on T1-weighted gadolinium enhanced MRI or contrast-enhanced CT) or leptomeningeal metastasis with positive CSF cytology study.
3. Patient whose brain parenchymal metastatic tumors either progress after WBRT, develop new lesions after WBRT, or CNS metastatic tumor do not response to WBRT according to image study 3 months after treatment. Patients with leptomeningeal metastasis does not necessarily need whole brain radiotherapy before enrollment.
4. Patients with Her2/neu overexpression or amplification will be allowed but will be informed about other available treatment options such as lapatinib plus capecitabine.
5. Patients must have adequate organ and marrow reserve measured within 14 days prior to randomization as defined below:

   * Absolute neutrophil count ≧1,000/mcL
   * Platelets ≧75,000/mcL
   * Total bilirubin ≦ 1.5 X upper normal limit
   * AST(SGOT)/ALT(SGPT) ≦ 2.5 X upper normal limit; for patients with liver metastases AST(SGOT)/ALT(SGPT) ≦ 5 X is allowed
   * Serum creatinine ≦ upper normal limit or creatinine clearance ≧50ml/min
   * Hemoglobin≧8.0 gm/dL
   * PTT ≦ upper normal limit; INR ≦ 1.5
   * Proteinuria ≤ 1+, if > 1+, urine protein must be ≦ 1 g/24 hours
6. Patient age 18 to 75 years
7. Patient's life expectancy is more than 2 months
8. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0, 1, 2 or 3
9. All women of childbearing potential must have a negative pregnancy test obtained within 72 hours before starting therapy
10. Patients with reproductive potential must use effective contraception (hormone or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 2 months after the completion of therapy
11. Patients (or a surrogate) must be able to comply with study procedures and sign informed consent

Exclusion criteria:

1. Prior therapy with bevacizumab, sorafenib, sunitinib, or other VEGF pathway-targeted therapy
2. Patients whose CNS metastasis progressed or developed during prior cisplatin treatment
3. History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
4. History of thrombotic disorders
5. Active gastrointestinal bleeding
6. Patients with a history of self-reported intra-cranial hemorrhage
7. Patients with clinical signs or symptoms of gastrointestinal obstruction and who require parenteral hydration and/or nutrition because of obstruction
8. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of first dose of bevacizumab
9. Clinically significant peripheral artery disease
10. Arterial thromboembolic event within the past 6 months, including transient ischemic attack, cerebrovascular accident, unstable angina, or myocardial infarction
11. History of gross hemoptysis (i.e. ≥ 1 teaspoon of bright red blood)
12. Other malignancy within 5 years except cured basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
13. Psychiatric illness or social situation that would preclude study compliance
14. Serious non-healing wound, ulcer, or bone fracture
15. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment
16. Prior minor surgery or needle biopsies within 7 days
17. Concurrent chronic daily aspirin (> 325 mg/day), dipyridamole, ticlopidine, clopidogrel, cilostazol, non-steroidal anti-inflammatory agents known to inhibit platelet function
18. Concurrent therapeutic anticoagulation, but prophylactic anti-coagulation of venous access devices is allowed
19. History of allergic reaction to compounds of similar chemical composition to the study drugs
20. Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Response rate of central nervous system (CNS) metastasis | 1 year
  The response criteria for brain parenchymal metastasis is measured according to the volumetric response criteria with modification. CNS lesion(s) which have a ≧ 50% volumetric reduction of in the absence of progressive neurologic signs and symptoms will be considered as responsive.
  The response criteria for leptomeningeal metastasis is defined as disappearance of carcinoma cells of three consecutive cytology examination of cerebrospinal fluid (CSF) after chemotherapy. For patients with both brain and leptomeningeal metastases, both criteria need to be met to be considered as responsive.

SECONDARY OUTCOMES:
Number of participants with adverse events | Baseline to until one month after last course of chemotherapy protocol treatment
  To observe the toxicity profile of B-EP according to CTCAE 3.0
To evaluate the response rate of breast cancer patients with brain parenchymal metastasis after receiving B-EP | 1 year
  To use volumetric measurement by subtraction image of CT the tumor before and after contrast enhancement; assessed every 9 weeks until best response measured
To evaluate the response rate of breast cancer patients with leptomeningeal carcinomatosis after receiving B-EP | 1 year
  A response is defined as the CSF cytology examination turns from positive to negative. A confirmed response is defined as CSF cytology examination remains negative for two or three consecutive tests
To evaluate the response rate of extra-CNS lesions according to RECIST | 1 year
  To evaluate the response rate of extra-CNS lesions according to RECIST. Measure every 9 weeks until best response recorded
Vascular activity of brain metastatic tumors after bevacizumab treatment | 4 weeks
  vascular activity detected with dynamic contrast enhanced magnetic resonance imaging (DCE-MRI), measured before treatment, 24 hours after bevacizumab administration and end of 1st cycle of B-EP
Biomarkers in CSF and serum in patients with brain and/or leptomeningeal metastasis receiving B-EP | Before the start of treatment till the end of treatment (after 6 cycles or progression)
  Prognostic and predictive value of biomarkers in CSF or serum. Serum will be drawn before treatment, end of cycle one and end of 6 cycles of treatment or time of progression
Drug concentrations of etoposide and cisplatin | 12 weeks
  Drug concentrations of bevacizumab, etoposide in CSF, blood and CSF/blood ratio before and after B-EP treatment in cycle one and cycle two
Association between response of CNS metastasis and the history of prior exposure to cisplatin | 1 year
  To evaluate the response rate and duration of response of CNS metastasis regarding to prior exposure to cisplatin
Proton MR spectroscopy of metastatic brain tumor before and after B-EP treatment | 4 weeks
  To evaluate the characteristics of 1H-MRS of metastatic brain tumor before and after B-EP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Shen Lu, MD, PhD, Principal Investigator — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taipei City, Taiwan

REFERENCES:
- [Derived] Chen BB, Lu YS, Lin CH, Chen WW, Wu PF, Hsu CY, Yu CW, Wei SY, Cheng AL, Shih TT. A pilot study to determine the timing and effect of bevacizumab on vascular normalization of metastatic brain tumors in breast cancer. BMC Cancer. 2016 Jul 13;16:466. doi: 10.1186/s12885-016-2494-8. PMID 27412562
- [Derived] Wu PF, Lin CH, Kuo CH, Chen WW, Yeh DC, Liao HW, Huang SM, Cheng AL, Lu YS. A pilot study of bevacizumab combined with etoposide and cisplatin in breast cancer patients with leptomeningeal carcinomatosis. BMC Cancer. 2015 Apr 17;15:299. doi: 10.1186/s12885-015-1290-1. PMID 25928457